CLINICAL TRIAL: NCT07131189
Title: A Phase I, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-Tumor Activity of FL115 Monotherapy in Subjects With Unresectable Locally Advanced or Metastatic Solid Tumors, Including Dose Escalation and Cohort Expansion
Brief Title: A Study of FL115 Monotherapy in Unresectable or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Forlong Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL115-102
Record Dates: First submitted 2025-07-21; First posted 2025-08-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced/Metastatic Solid Tumors

STUDY DESIGN:
Intervention Model Description: Open-label, Multicenter, Dose escalation and Expansion part
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Single Arm (Experimental)
  Interventions: Drug: FL115

INTERVENTIONS:
Drug: FL115 — FL115 is a novel long-acting IL-15 agonist designed as a fusion protein with a mutated IL-15 structure (IL-15[N72D]/IL-15Rα-sFc).

SUMMARY:
This is a Phase 1, open-label, multicenter clinical study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of FL115 administered as monotherapy in subjects with unresectable locally advanced or metastatic solid tumors. The study consists of a dose escalation phase followed by a dose expansion phase to further characterize the safety profile and clinical activity at the recommended dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older and up to 80 years old.
2. Subjects with locally advanced or metastatic solid tumors that have been pathologically or cytologically confirmed and have failed all standard treatments, currently have no standard treatment options, or are not suitable for standard treatment.
3. With at least one measurable lesion (according to RECIST v1.1).
4. ECOG score: 0 - 1.
5. Expected survival period ≥ 12 weeks (judged by the investigator).
6. Sufficient organ function.
7. Voluntary written informed consent and agree to comply with all protocol-specified procedures and follow-up evaluations.
8. Fertile subjects (male and female) and their partners agree to use acceptable, investigator-approved contraception during the study-required period.

Exclusion Criteria:

If any of the following criteria are met, the subjects will be excluded from the study:

1. History of previous anti-tumor treatment:

   1. Previous use of IL-2 or IL-15 agonists, including but not limited to rhIL-15 (NCI), ALT-803 (ALTOR), NKTR-214 (Nektar).
   2. Received any anti-tumor investigational or approved drug, biologic, or endocrine immunotherapy (except HRT, oral contraceptives, testosterone, ADT for prostate cancer, or endocrine therapy for breast cancer) within 4 weeks before first dose; or received >30Gy non-thoracic radiotherapy or within 4 weeks or >30Gy lung radiotherapy within 8 weeks; or ≤30Gy palliative radiotherapy within 14 days before first dose.
   3. Within 2 weeks before the first administration of the study drug, received traditional Chinese medicine for anti-tumor indications.
   4. Subjects who received oral fluoropyrimidines or small-molecule targeted therapies discontinued the treatment ≤2 weeks or 5 half-lives (whichever is longer) prior to the first dose of the study drug.
   5. Subjects who received mitomycin C or nitrosourea treatment discontinued the medication ≤6 weeks prior to the first dose of the study drug.
2. History of other previous treatments and toxicity recovery:

   1. Known or suspected allergies to FL115 and its excipients; known history of grade 3-4 allergic reactions to interleukin treatment or other fusion proteins.
   2. Known allergies to indomethacin, acetaminophen, diphenhydramine, ranitidine, cimetidine and/or famotidine.
   3. Received systemic immunosuppressants within 4 weeks before first dose, except for: ≤10 mg/day prednisone-equivalent, local/inhaled/nasal steroids, ≤7.5 mg/day for adrenal replacement, or one-time use for contrast allergy before imaging.d) .
   4. Received treatment with granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), thrombopoietic agents (e.g., thrombopoietin [TPO], romiplostim, eltrombopag), or erythropoiesis-stimulating agents (e.g., erythropoietin [EPO]) within 14 days prior to screening.
   5. History of allogeneic organ or PBSC/bone marrow transplant.
   6. Received live viral vaccine within 4 weeks before first dose.
   7. Prior ≥Grade 3 or treatment-discontinuing irAEs, except for hypothyroidism, type 1 diabetes, or mild skin irAEs (excluding SJS, TEN, or severe dermatitis).
   8. Before first dose, all AEs from prior anti-tumor therapy have not resolved to baseline or ≤Grade 1 (per NCI CTCAE v5.0). Exceptions: hair loss (any grade) and ≤Grade 2 peripheral neuropathy are allowed; other ≤Grade 2 AEs may be allowed if deemed acceptable by the investigator and inclusion should be discussed with the sponsor's medical monitor.
3. Past medical history and surgical history:

   1. Malignant tumors of the blood system (such as acute lymphocytic leukemia, acute myeloid leukemia, myelodysplastic syndrome, chronic lymphocytic leukemia, chronic myeloid leukemia, non-Hodgkin's lymphoma, Hodgkin's lymphoma, and multiple myeloma).
   2. Subjects with active central nervous system (CNS) metastatic lesions or meningeal metastasis. Exception: Asymptomatic subjects with CNS metastatic tumors if the clinical condition is controlled.
   3. Subjects who had other malignant tumors within 2 years before screening. Subjects with curable local tumors (such as basal or squamous cell skin cancer, cervical or breast carcinoma in situ), can be included after clear cure.
   4. Have active autoimmune diseases or a history of autoimmune diseases requiring systemic steroids or immunosuppressants, such as rheumatoid arthritis, lupus, Wegener's granulomatosis, Sjogren's syndrome, IBD, multiple sclerosis, myasthenia gravis, myositis, autoimmune hepatitis, vasculitis, immune thrombocytopenia, autoimmune hemolytic anemia, or glomerulonephritis.

Exception: subjects with well-controlled endocrine disorders treated with HRT (e.g., hypothyroidism, type 1 diabetes).

e) Subjects had any of the following pulmonary toxic reactions/diseases in the past:

1. Significantly clinically significant severe pulmonary-specific diseases, including but not limited to: pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease, history of idiopathic pulmonary fibrosis, organizing pneumonia (such as obliterative bronchiolitis), history of drug-induced pneumonia;
2. Active interstitial lung disease (ILD) or interstitial pneumonia; history of requiring hormone or other immunosuppressant treatment for ILD or (non-infectious) pneumonia;
3. Found by history or CT examination that there was active tuberculosis infection within 1 year before enrollment or more than 1 year ago with no regular treatment; f) Judged by the investigator to have uncontrollable pleural effusion, pericardial effusion, or peritoneal effusion.

   g) Have a significant clinical history of cardiovascular diseases. h) Underwent major surgery within 4 weeks prior to signing the informed consent form.
4. Infectious Disease History:

   1. Severe infections within 4 weeks before first dose.
   2. Any history of confirmed active HBV, HCV, HIV, or active tuberculosis infection.
5. Other Conditions:

   1. Pregnant or breastfeeding women.
   2. Known, documented, or suspected substance abuse. Exceptions: Prescribed opioids for pain control or other investigator-approved, medically justified cases (pending sponsor medical lead agreement).
   3. Any other conditions deemed by the investigator to render the subject unsuitable for participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerabilty | through study completion, an average of 8months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
MTD | up to 18 months
  Maximal Tolerance Dose
RP2D | up to 18 months
  Recommended Phase II Dose

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shandong Cancer Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No
Our research is based on earlier studies and there is a high degree of uncertainty. We will consider sharing the results only after we have obtained sufficient data.